CLINICAL TRIAL: NCT04249414
Title: Post-hoc Analysis of Regional Pulmonary Perfusion and Hemodynamic Parameters Measured by Electrical Impedance Tomography
Status: Suspended | Type: Observational
Why Stopped: Due to a lack of resources (human and financial), it is currently unclear if the study will be counducted.
Sponsor: Drägerwerk AG & Co. KGaA (Industry)
Collaborators: University of Göttingen (Other); Prof. Dr. med. Imhoff (Unknown)
Responsible Party: Sponsor
Other Study IDs: PV500PERF
Record Dates: First submitted 2020-01-27; First posted 2020-01-31 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Mechanical Ventilation; Ventilation Perfusion Mismatch
Keywords: Ventilation Monitoring; Electrical Impedance Tomography; Perfusion Monitoring; Hemodynamic Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PulmoVista 500 — Monitoring of Ventilation and Perfusion with the PulmoVista 500 during clinical routine.
  No medical interventions required

SUMMARY:
Define the capability and reliability of the PulmoVista® 500 (PV500) to detect changes in global and regional ventilation and perfusion.

DETAILED DESCRIPTION:
The results of this study will help defining the capability and reliability of PulmoVista® 500 (PV500) to detect changes in both global and regional ventilation and perfusion. As this is a non-invasive, observational trial, neither a positive nor a negative impact on the actual study participants is expected. The results will, however, improve the knowledge about the electrical impedance tomography (EIT) technology and thus aid the use of this technology for the benefit of future patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years
* Mandatorily ventilated intensive-care patients with impairment in oxygenation (P/F ratio < 300 at PEEP ≥ 5) ventilated at a positive end-expiratory pressure (PEEP) not exceeding 10 mbar and an fraction of inspired oxygen (FiO2) chosen, such that pulse oximetry is sensitive towards arterial oxygen pressure (PaO2) changes.
* Expected ventilation time >48h
* Existing central venous and arterial access
* Chest circumference 70 - 150 cm
* Mandatory mechanical ventilation (patients without spontaneous efforts)
* Serum levels of sodium and chloride within normal range
* Cardiac output monitoring in place (PICCO)

Exclusion Criteria:

* Contraindication to central venous injection of 5 % sodium chloride (NaCl) (e.g. elevated Na+ and/or Cl- concentration: Na+ should not exceed 150 mmol/l, Chloride should not exceed 115 mmol/l, known hypernatremia, known high serum osmolality)
* Contraindications of PulmoVista 500:

  * Patients with pacemakers, defibrillators or other electrically active implants
  * Patients with damaged skin or impaired skin contact of the electrodes due to wound dressings
  * Patients where the attachment of the patient belt could pose a risk to the patient, e.g. patients with spinal lesions or fractures
  * Patients with uncontrolled body movements
  * Extremely obese patients (BMI>50)
  * Patients during pregnancy
  * Patients with massive lung edema
  * Use during electricity-based therapies, such as electrosurgery or electrocautery
  * Use in the presence of strong magnetic fields
  * Use in conjunction with other bioimpedance measurement devices
* Infection or colonization with multi-resistant pathogens that require isolation of the patient (e.g. MRSA)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the ICU who are mandatorily ventilated for at least 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Assess regional distribution of pulmonary perfusion | within 24 hours
  The capability of PulmoVista® 500 for assessing regional distribution of pulmonary perfusion based on pulsatility signals and based on indicator dilution and changes at different points in time during varying states of regional ventilation will be evaluated.

SECONDARY OUTCOMES:
Assess hemodynamic parameter cardiac output | within 24 hours
  The capability of PulmoVista® 500 for assessing cardiac output (relative values compared to reference given in l/min) will be explored.
Assess hemodynamic parameter heart rate | within 24 hours
  The capability of PulmoVista® 500 for assessing heart rate (1/min) will be explored.
Assess hemodynamic parameter stroke volume variability | within 24 hours
  The capability of PulmoVista® 500 for assessing stroke volume variability (relative value in % for 30 seconds compared to reference given in ml) will be explored.
Assess oxygenation status | within 24 hours
  The capability PulmoVista® 500 for assessing the oxygenation status from both the regional distribution of alveolar ventilation and the regional distribution of pulmonary perfusion will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Onnen Mörer, Prof. Dr., Principal Investigator — Centre of Anaesthesiology University Medical Center Göttingen; Michael Quintel, Prof. Dr., Study Director — Centre of Anaesthesiology University Medical Center Göttingen
Locations (1):
- University Medical Center Göttingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No